CLINICAL TRIAL: NCT01238185
Title: Oral Topical Cyclooxygenase Inhibitor (Aspirin) Mouthwash for Treatment of Oral Dysplasia
Brief Title: Aspirin Mouthwash in Treating Patients With Oral Leukoplakia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Institute of Head and Neck Studies and Education, United Kingdom (Other)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: INHANSE-ASPOD; CDR0000688122 (Registry Identifier: PDQ (Physician Data Query)); ISRCTN31503555 (Registry Identifier: ISRCTN (International Standard Randomised Controlled Trial Number Register)); EU-21083
Record Dates: First submitted 2010-11-09; First posted 2010-11-10 (Estimated); Last update posted 2013-08-12 (Estimated); Status verified 2010-11

CONDITIONS: Precancerous Condition
Keywords: oral leukoplakia
MeSH Terms: conditions — Precancerous Conditions; Leukoplakia, Oral | interventions — Aspirin; Gene Expression Profiling; Biopsy

INTERVENTIONS:
Drug: acetylsalicylic acid
Genetic: gene expression analysis
Genetic: protein expression analysis
Other: laboratory biomarker analysis
Other: questionnaire administration
Procedure: biopsy

SUMMARY:
RATIONALE: Aspirin mouthwash may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

PURPOSE: This phase I trial is studying the side effects and best dose of aspirin mouthwash in treating patients with oral leukoplakia.

DETAILED DESCRIPTION:
OBJECTIVES:

* To determine if oral topical acetylsalicylic acid mouthwash achieves modulation of COX-1, COX-2, and prostaglandin in oral dysplasia tissues in patients with oral leukoplakia.
* To determine if this drug achieves alteration of histopathology and gene and protein expression in tissue.
* To determine if this drug achieves aspirin-induced tissue changes relating to altered tumor biology.
* To assess local and general tolerability and safety of this drug in these patients.

OUTLINE: All patients undergo tissue biopsy for histological diagnosis. Patients without a histological diagnosis of precancerous oral dysplasia undergo routine follow-up. Patients with a histological diagnosis of precancerous oral dysplasia are sequentially allocated to 1 of 4 treatment groups.

* Group 1: Patients receive acetylsalicylic acid mouthwash (one 75 mg tablet dissolved in 250 mL of water) twice daily for 4-6 weeks, gargling for 60 seconds then expectorate it fully, before planned definitive surgical excision.
* Group 2: Patients receive acetylsalicylic acid mouthwash (two 75 mg tablets of acetylsalicylic acid dissolved in 250 mL of water) twice daily for 4-6 weeks, gargling for 60 seconds then expectorate it fully, before planned definitive surgical excision.
* Group 3: Patients receive acetylsalicylic acid mouthwash (one 300 mg tablet of acetylsalicylic acid dissolved in 250 mL of water) twice daily for 4-6 weeks, gargling for 60 seconds then expectorate it fully, before planned definitive surgical excision.
* Group 4: Patients receive acetylsalicylic acid mouthwash (one 300 mg tablet of acetylsalicylic acid dissolved in 250 mL of water) three times daily for 4-6 weeks, gargling for 60 seconds then expectorate it fully, before planned definitive surgical excision.

At the time of definitive surgical excision, the patient is asked to gargle with the last dose of acetylsalicylic acid mouthwash just before being anesthetized. A small biopsy of the dysplasia lesion is taken and examined for immediate effects of the acetylsalicylic acid mouthwash on the dysplasia lesion. The surgically excised tissue is treated in the same way as the initial biopsy tissue (i.e., half being used for routine histology to confirm the diagnosis and the other half for research purposes). Tissue samples are analyzed via enzyme immunosorbent assay, qRT-PCR, immunoblotting, ELISA, immunohistochemistry, gene array analysis, and microvessel density analysis.

Patients complete a questionnaire assessing local and general tolerability as well as adverse effects during the period of use of the mouthwash.

After completion of study treatment, patients are followed periodically.

Peer Reviewed and Funded or Endorsed by Cancer Research UK

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Clinically diagnosed oral leukoplakia requiring a tissue biopsy for histological diagnosis
* Attending the outpatient clinic

PATIENT CHARACTERISTICS:

* Not nursing
* No known or suspected sensitivity to aspirin or other nonsteroidal anti-inflammatory drugs
* No diagnosis of asthma or angioedema
* No contraindications, including any of the following:

  * Active peptic ulceration or a history of peptic ulceration
  * Hemophilia or a history of bleeding disorders
  * Gout or a history of gout

PRIOR CONCURRENT THERAPY:

* No concurrent regular use of aspirin for heart disease or other reasons
* No other concurrent nonsteroidal anti-inflammatory drugs

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2010-02; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
PGE2 levels as assessed by enzyme immunosorbent assay
COX-1 and COX-2 mRNA as assessed by qRT-PCR
COX-1 and COX-2 protein expression as assessed by immunohistochemistry and quantified by immunoblotting to determine whether COX inhibition in oral dysplasia tissues is actually possible by use of the mouthwash formulation

SECONDARY OUTCOMES:
Comparison of WHO histological grade and clinical size of dysplastic lesions before and after treatment and assessment of proliferating cell nuclear antigen
Tolerability and possible oral and other adverse effects using a questionnaire
VEGF mRNA expression as assessed by qRT-PCR
Protein expression as assessed by ELISA and immunohistochemistry for VEGFA
Global gene response of dysplastic tissue as assessed by Affymetrix gene expression microarrays

CONTACTS AND LOCATIONS:
Overall Officials: Hisham Mehanna, MD, Principal Investigator — Institute of Head and Neck Studies and Education, United Kingdom
Locations (2):
- United Kingdom (2):
  - University of Birmingham, Birmingham, England
  - Institute of Head and Neck Studies and Education, Coventry, England